CLINICAL TRIAL: NCT07153341
Title: A Pre-Post Trial Evaluating the Supporting Transitions and Empowering Preferences (STEP) Decision Support Intervention for Long-Term Care Residents Facing Hospital Transfer Decisions During Acute Health Crises
Brief Title: Evaluation of the STEP Intervention for Long-Term Care Residents Facing Hospital Transfer Decisions
Acronym: STEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: M16-25-017; 478736 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-08-19; First posted 2025-09-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: LTC-to-hospital Transfer Decision-making
Keywords: long-term care; hospital transfers; acute health events; decision-making in older adults; resident-centred care; substitute decision-makers; frailty; cognitive impairment; shared decision-making; avoidable hospitalizations; transitional care; decision aid; health decision support; decision coaching; pre-post intervention study; healthcare quality improvement; decisional conflict; decisional regret
MeSH Terms: conditions — Frailty; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This trial uses a pre-post evaluation design at two LTC sites. All participants receive the same intervention (the STEP tool), with no comparison group or randomization to different arms. Outcomes are compared before and after the intervention within the same group (resident-care partner dyads and nurses).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STEP Intervention (Experimental): Participants (resident-care partner dyads) in this arm will receive the STEP intervention. STEP is a decision aid designed to support shared decision-making about whether to transfer to hospital or remain in LTC during acute health events. It includes an educational booklet, a structured decision aid, and a staff phone script used at three points in the resident's care journey: (1) upon LTC admission, (2) during annual care conferences, and (3) at the time of an acute medical event. LTC nurses will receive training to deliver the STEP tool and support residents and care partners in making informed, values-based transition decisions.
  Interventions: Behavioral: STEP Decision Support Toolkit

INTERVENTIONS:
Behavioral: STEP Decision Support Toolkit — The STEP toolkit includes (1) an educational booklet provided upon admission and annually, (2) condition-specific decision aids addressing common clinical scenarios, and (3) structured phone scripts for staff. STEP empowers residents and care partners to actively engage in decision-making, promotes care aligned with personal values, and supports staff in facilitating advance care planning to reduce unnecessary or complex transitions.

SUMMARY:
This trial will evaluate whether the Supporting Transitions and Empowering Preferences (STEP) toolkit can improve decision-making about hospital transfers in long-term care residents and their substitute decision-makers and enhance decision self-efficacy in nursing staff.

The trial will answer the questions:

* Does the STEP tool reduce decisional conflict in residents and care partners at the time of transfer decisions?
* Does it improve nurse self-efficacy related to hospital transfer decisions?

Participants will:

* Use the STEP tool during key moments of care planning (admission, care conferences, and acute events)
* Complete a short survey measuring their decisional conflict
* Be supported by trained nurses who use STEP to guide hospital transfer discussions

Researchers will compare data collected before and after the STEP tool is implemented at two long-term care homes to see if it improves shared decision-making related to hospital transfers by reducing decisional conflict.

DETAILED DESCRIPTION:
Background and Rationale: Transitions from long-term care (LTC) to hospital are complex and can offer both benefits and challenges to residents and care partners. While LTC-to-hospital transitions can improve health outcomes, particularly during acute deterioration, evidence also indicates that these transitions may disrupt continuity of care, increase stress, and misalign resident needs with hospital protocols. Nearly fifty percent of LTC residents in Canada experience hospital transitions annually, with approximately forty percent considered avoidable. Risks include non-evidence-based care, safety concerns, unnecessary interventions, and increased mortality rates. Transition decisions are influenced by residents' health status, medico-legal concerns, staff workload, and care partners' confidence in LTC care. These decisions are often reactive and shaped by unequal power dynamics rather than proactive, collaborative planning.

Given these challenges, and limitations in current monitoring systems such as the Minimum Data Set assessments, there is a critical need for a decision aid that supports informed, resident-centered planning. The Supporting Transitions and Empowering Preferences (STEP) tool was developed through interviews, co-design sessions, document analysis, and stakeholder engagement.

Objectives Primary Objective: Evaluate the impact of STEP on decisional conflict among residents and care partners.

Secondary Objective: Examine the effect of STEP on nurses' self-efficacy as decision coaches at the time of transition decisions.

Trial Design and Study Setting: A pre-post evaluation will be conducted at two LTC sites (Perley Health and Bruyère Health Saint-Louis LTC) to assess STEP's ability to support resident-care partner dyads in making hospital transition decisions. STEP will be implemented simultaneously at both sites.

Study Overview: Data will be collected for six months pre-intervention or until the target sample size is reached (n=100), followed by the intervention period. Nurses, nurse practitioners, social service workers, and physicians will receive STEP training, with designated champions supporting implementation. Data will be collected at three points: after intake/admission meetings, after care conferences, and after acute events in which a transfer is considered.

Vanguard Phase Implementation: An initial vanguard phase involving approximately ten residents over four to six weeks will test feasibility, refine recruitment, and assess staff comfort before broader rollout.

Description of the Intervention (Overview): The STEP intervention includes three resources: (1) an educational booklet about transition decisions, (2) a structured decision aid, and (3) a phone script for nursing staff calling substitute decision-makers at the time of a transfer decision. Staff will be trained on the use of these resources with sessions scheduled to accommodate different shifts. STEP will be introduced at admission (educational booklet), reviewed at post-admission or annual care conferences (booklet + decision aid), and used during acute health events (decision aid + phone script) to guide structured conversations about hospital transfer decisions.

Monitoring Fidelity: Implementation fidelity will be monitored through nurse logs, informal discussions, and champion reports, assessing feasibility, acceptability, and adherence.

Data Collection Procedures (Overview): Dyads will be identified through care reports and hospital transfer notifications, with eligibility verified prior to consent. Data will be collected using secure REDCap software. For nurses, care conference and physician call notes will be reviewed to identify eligible cases. Surveys and brief interviews will assess experiences, confidence, and barriers to STEP use.

Analysis: Analyses will follow an intention-to-treat approach using Generalized Estimating Equations for repeated measures. Differences between groups will be examined using t-tests or chi-squared tests. Missing data will be minimized through follow-up; cases lost after three unsuccessful contact attempts will be excluded from analysis.

ELIGIBILITY:
Inclusion Criteria

Residents-care partner dyads:

* Must be residents of either Perley Health or Bruyère Health Saint-Louis LTC home.
* Residents must be 55 years of age or older.
* Must be able to communicate in French or English.

Both members of the dyad will be included where applicable. For dyads in which residents do not have the capacity to participate, inclusion will occur through the involvement of their substitute decision-maker (e.g., power of attorney for personal care).

LTC staff:

* Must be a nurse, nurse practitioner, social service worker or physician actively involved in care planning, annual conferences, or managing acute health events at Perley Health or Bruyère Health.
* Must have been employed at the LTC home for at least 6 months to ensure familiarity with the care environment and residents.
* Must play a role in facilitating discussions, providing clinical input (where applicable), or guiding decision-making processes related to hospital transitions or acute care management.
* Must be able to communicate in French or English.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-04 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict | Administered by Research Assistant 1-6 weeks after a transition decision.
  Measured using the Decisional Conflict Scale (16 items; each rated on a 5-point scale; standardized total score 0-100, with higher scores indicating greater decisional conflict and worse decision-making outcomes).

SECONDARY OUTCOMES:
Decision Self-Efficacy | Administered by Research Assistant 1-6 weeks after a transition decision and periodically thereafter.
  Measured using the Decision Self-Efficacy Scale (11 items; each rated 0-4, standardized to a 0-100 score, with higher scores indicating greater decision self-efficacy and better outcomes).
Transition Rate | Measured continuously during the 6 months pre-intervention and 6 months post-intervention periods.
  Measured as the rate of hospital transitions during the pre- and post-intervention periods, including: (1) total number of transitions documented in electronic medical records; (2) avoidable transitions, defined as transitions for conditions that could have been managed in the LTC home (e.g., non-critical infections, falls without significant injury); and (3) repeat transitions, defined as multiple transitions experienced by the same resident within a 6-month period.
Resident Health Outcomes Post-Transition | Measured continuously during the 6 months pre-intervention and 6 months post-intervention periods.
  Measured as the rate of rehospitalizations within 30 days of discharge among residents who experienced a hospital transition. This outcome will be assessed using electronic medical records, contingent on resident consent and feasibility of participant identification. Higher rates indicate worse health outcomes.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Bruyère Health Saint-Louis Long-Term Care, Ottawa, Ontario
  - Perley Health, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No
Given the small sample size, the sensitive nature of data collected in long-term care settings, and the potential risk of participant re-identification, we do not plan to share IPD publicly. However, IPD may be shared on a case-by-case basis in response to reasonable, ethically approved requests. Aggregate results will be disseminated through publications and presentations.

REFERENCES:
- [Background] Tappen RM, Elkins D, Worch S, Weglinski M. Modes of Decision Making Used by Nursing Home Residents and Their Families When Confronted With Potential Hospital Readmission. Res Gerontol Nurs. 2016 Nov 1;9(6):288-299. doi: 10.3928/19404921-20160920-01. Epub 2016 Sep 27. PMID 27665753
- [Background] Marincowitz C, Preston L, Cantrell A, Tonkins M, Sabir L, Mason S. What influences decisions to transfer older care-home residents to the emergency department? A synthesis of qualitative reviews. Age Ageing. 2022 Nov 2;51(11):afac257. doi: 10.1093/ageing/afac257. PMID 36413591
- [Background] Gruneir A, Bronskill SE, Newman A, Bell CM, Gozdyra P, Anderson GM, Rochon PA. Variation in Emergency Department Transfer Rates from Nursing Homes in Ontario, Canada. Healthc Policy. 2016 Nov;12(2):76-88. PMID 28032826
- [Background] Gruneir A, Anderson GM, Rochon PA, Bronskill S. Transitions in long-term care and potential implications for quality reporting in Ontario, Canada. J Am Med Dir Assoc. 2010 Nov;11(9):629-35. doi: 10.1016/j.jamda.2010.07.007. PMID 21029997
- [Background] Cummings GG, McLane P, Reid RC, Tate K, Cooper SL, Rowe BH, Estabrooks CA, Cummings GE, Abel SL, Lee JS, Robinson CA, Wagg A. Fractured Care: A Window Into Emergency Transitions in Care for LTC Residents With Complex Health Needs. J Aging Health. 2020 Mar;32(3-4):119-133. doi: 10.1177/0898264318808908. Epub 2018 Nov 15. PMID 30442040
- [Background] Abraham S, Menec V. Transitions Between Care Settings at the End of Life Among Older Homecare Recipients: A Population-Based Study. Gerontol Geriatr Med. 2016 Dec 15;2:2333721416684400. doi: 10.1177/2333721416684400. eCollection 2016 Jan-Dec. PMID 28680944
- [Background] Menard A, Singh Y, Adams M, Bai JQA, Kobewka D, MacLeod KK. "We Didn't Ask to Be Sick:" Equipping Residents and Care Partners for Transitions From Long-Term Care to Hospital. J Am Geriatr Soc. 2025 Aug;73(8):2410-2421. doi: 10.1111/jgs.19535. Epub 2025 May 30. PMID 40444661
- [Background] Menard A, Konikoff L, Adams M, Singh Y, Scott MM, Yin CY, Kimura M, Kobewka D, Fung C, Isenberg SR, Kaasalainen S, Kierulf J, Molnar F, Shamon S, Wilson K, Kehoe MacLeod K; Ottawa Hospital Research Institute and Bruyere Health Research Institute. Supporting resident-centred decision-making about transitions from long-term care homes to hospital: a qualitative study protocol. BMJ Open. 2024 Nov 29;14(11):e086748. doi: 10.1136/bmjopen-2024-086748. PMID 39615892